CLINICAL TRIAL: NCT00104546
Title: Vitamin K Injection Treatment for Primary Dysmenorrhea: A Controlled Pilot Study
Brief Title: Vitamin K Injections for the Treatment of Painful Menstruation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT001957 (NIH)
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; Acupuncture; Vitamin K; Medicine, Chinese Traditional; Women; Menstruation; Pain, Menstrual; China
MeSH Terms: conditions — Dysmenorrhea

INTERVENTIONS:
Procedure: Acupuncture point injection of vitamin K

SUMMARY:
The purpose of this study is to test the feasibility and effectiveness of vitamin K injections into certain body parts for the treatment of painful menstruation.

DETAILED DESCRIPTION:
Painful menstruation, also known as dysmenorrhea, is a common problem affecting a significant percentage of women. In the United States and Europe, nonsteroidal anti-inflammatory drugs (NSAIDs) and oral contraceptives are the most commonly prescribed treatments for this condition. However, in China, oral contraceptives are not commonly prescribed for unmarried women. Acu-injection, a procedure involving the injection of vitamin K into acupuncture points, has become standard treatment for dysmenorrhea at many Chinese health care facilities. This trial will assess the willingness of young Chinese women to participate in an acu-injection trial, explore the utility of pain measurements after injection, and determine the effectiveness of the injections. This study will also help in planning larger acu-injection clinical trials.

This study will last for five menstrual cycles. Participants will be randomly assigned to one of three groups. Group 1 participants will receive a vitamin K3 injection in an acupuncture point of both legs and a saline injection in the right buttock. Group 2 participants will receive a saline injection in an acupuncture point of both legs and a saline injection in the right buttock. Group 3 participants will receive a saline injection in a pseudo-acupuncture point of both legs and a vitamin K3 injection in the right buttock. Injections will be administered one time during the first 2 days of the first menstrual cycle for participants who are experiencing menstrual pain. Participants will record their level of menstrual pain before injection and at 2, 5, 30 and 60 minutes after the injections. Participants who do not respond to or are not satisfied with the acu-injection treatment will be offered either Chinese herbal medicine or NSAIDs within 1 hour of the injection. After the injection visit, participants will be asked to complete questionnaires about any menstrual pain or side effects they may be experiencing for five subsequent menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* Dysmenorrhea for at least 6 months prior to study entry
* Have never been pregnant or have given birth
* Mandarin Chinese or Shanghainese speaking
* Regular menstrual cycles for at least 6 months prior to diagnosis of dysmenorrhea
* Has a working home phone or cellular phone
* Willing to disclose address
* Intends to stay in the area during the study
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Dysmenorrhea due to any suspected or recognized causes
* Current use of hormonal contraceptives or an intrauterine device
* History of abdominal surgery
* Other concomitant therapy for acute or chronic pain
* Anticoagulant drugs
* Vitamin K acu-injections at leg acupuncture points prior to study entry
* Intolerance to NSAIDs
* Known allergy to vitamin K

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36
Dates: Start 2004-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Intensity of menstrual pain before and 2, 5, 30, and 60 minutes after treatment by a 10 point Visual Analog Scale (VAS)
presence and severity of recurrences of menstrual pain pre- and post-treatment and in 5 subsequent cycles after therapy
Cox retrospective symptom scale
Moos score

CONTACTS AND LOCATIONS:
Overall Officials: Fredi Kronenberg, PhD, Principal Investigator — Columbia University
Locations (1):
- Menstrual Disorder Clinic of the OBS/GYN Hospital of Fudan University, Shanghai, China

REFERENCES:
- [Derived] Wade C, Wang L, Zhao WJ, Cardini F, Kronenberg F, Gui SQ, Ying Z, Zhao NQ, Chao MT, Yu J. Acupuncture point injection treatment of primary dysmenorrhoea: a randomised, double blind, controlled study. BMJ Open. 2016 Jan 5;6(1):e008166. doi: 10.1136/bmjopen-2015-008166. PMID 26733563